CLINICAL TRIAL: NCT04344795
Title: Phase 1a/1b Open Label Dose-escalation and Expansion Study of TPST-1495 as a Single Agent and in Combination With Pembrolizumab in Subjects With Solid Tumors
Brief Title: Phase 1a/1b Study of TPST-1495 as a Single Agent and in Combination With Pembrolizumab in Subjects With Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tempest Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: TPST-1495-001
Record Dates: First submitted 2020-04-07; First posted 2020-04-14 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Solid Tumor; Colorectal Cancer; Non Small Cell Lung Cancer; Squamous Cell Carcinoma of Head and Neck; Urothelial Carcinoma; Endometrial Cancer; Gastroesophageal Junction Adenocarcinoma; Gastric Adenocarcinoma; Solid Tumors With PIK3Ca Mutation
Keywords: TPST-1495; EP2 antagonist; EP4 antagonist; prostaglandin E2 (PGE2); pembrolizumab; PIK3Ca mutation
MeSH Terms: conditions — Colorectal Neoplasms; Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck; Carcinoma, Transitional Cell; Endometrial Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: open-label dose escalation, schedule and dose optimization, and dose expansion
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- TPST-1495 monotherapy dose escalation (Experimental): Subjects will receive escalating doses of TPST-1495 administered orally twice daily until maximum tolerated dose is reached or until disease progression
  Interventions: Drug: TPST-1495 twice daily
- TPST-1495 monotherapy dose and schedule optimization (Experimental): Subjects will receive alternative TPST-1495 administration schedules until RP2D for the selected schedule is determined or until disease progression.
  Interventions: Drug: TPST-1495 once daily or on intermittent schedule
- TPST-1495 monotherapy dose expansion (Experimental): Subjects will receive selected dose regimen from dose and schedule optimization stage until disease progression
  Interventions: Drug: TPST-1495 once daily or on intermittent schedule
- TPST-1495 in combination with pembrolizumab dose and schedule optimization (Experimental): Subjects will receive alternative TPST-1495 administration schedules in combination with pembrolizumab until RP2D for the selected schedule is determined or until disease progression.
  Interventions: Drug: TPST-1495 once daily or on intermittent schedule; Drug: Pembrolizumab
- TPST-1495 in combination with pembrolizumab dose expansion (Experimental): Subjects will receive selected dose regimen from dose and schedule optimization stage until disease progression
  Interventions: Drug: TPST-1495 once daily or on intermittent schedule; Drug: Pembrolizumab

INTERVENTIONS:
Drug: TPST-1495 twice daily — TPST-1495 administered orally twice daily
  Arms: TPST-1495 monotherapy dose escalation
Drug: TPST-1495 once daily or on intermittent schedule — TPST-1495 administered orally once daily or on intermittent schedule
  Arms: TPST-1495 in combination with pembrolizumab dose and schedule optimization; TPST-1495 in combination with pembrolizumab dose expansion; TPST-1495 monotherapy dose and schedule optimization; TPST-1495 monotherapy dose expansion
Drug: Pembrolizumab — Pembrolizumab dosed per label recommendations
  Other Names: Keytruda
  Arms: TPST-1495 in combination with pembrolizumab dose and schedule optimization; TPST-1495 in combination with pembrolizumab dose expansion

SUMMARY:
This is a first-in-human Phase 1a/1b, multicenter, open-label, dose-escalation, dose and schedule optimization, and expansion study of TPST-1495 as a single agent and in combination with pembrolizumab to determine its maximum tolerated dose (MTD) and or recommended Phase 2 dose (RP2D), safety, tolerability, pharmacokinetics, pharmacodynamics and preliminary anti-tumor activity in subjects with advanced solid tumors. Subjects with all histologic types of solid tumors are eligible for the escalation and dose-finding portions of the study. However, the preferred tumor types for enrollment are colorectal cancer (CRC), non-small cell lung cancer (NSCLC), squamous cell carcinoma of the head and neck (SCCHN), urothelial cancer, endometrial cancer, and gastroesophageal junction (GEJ) or gastric adenocarcinoma. Enrollment in the expansion cohorts is limited to the following tumor types: endometrial, SCCHN, CRC, and a basket cohort in subjects selected for an activating mutation in PIK3Ca.

DETAILED DESCRIPTION:
This is a first-in-human Phase 1a/1b, multicenter, open-label, dose-escalation, dose and schedule optimization, and expansion study of TPST-1495 as a single agent and in combination with pembrolizumab to determine its MTD, safety, tolerability, pharmacokinetics (PD), pharmacodynamics (PK) and preliminary anti-tumor activity in subjects with advanced solid tumors. Subjects with all histologic types of solid tumors are eligible for the study. However, the preferred tumor types for enrollment are colorectal cancer (CRC), non-small cell lung cancer (NSCLC), squamous cell carcinoma of the head and neck (SCCHN), urothelial cancer, endometrial cancer, and gastroesophageal junction (GEJ) or gastric adenocarcinoma. Tumor prostaglandin production and downstream signaling in both tumor cells and other cell types, including immune suppressive cell population in the tumor microenvironment, is thought to be a principal driver of progression in each of these selected malignancies. To be eligible, subjects must have no remaining standard therapy known to confer clinical benefit.

The study is composed of 3 stages. The Dose-Escalation stage will determine the MTD of single-agent TPST-1495 administered twice a day (BID). The Schedule and Dose Optimization stage will evaluate alternative TPST-1495 single-agent administration schedules and determine an RP2D for the selected schedule. This arm will also evaluate TPST-1495 in combination with pembrolizumab. The Expansion stage will evaluate the activity of TPST-1495 as a single agent and in combination with pembrolizumab at the selected schedule and dose in disease-specific cohorts and in a basket cohort in subjects selected for an activating mutation in PIK3Ca.

ELIGIBILITY:
Subjects must meet all the following inclusion criteria to be eligible:

1. Subjects must have a histologically-confirmed malignancy that is metastatic or unresectable for which there is no remaining standard therapy known to confer clinical benefit. While all solid tumor types are eligible for the dose-escalation and dose-finding portions of the study, there is a preference to enroll patients with colorectal cancer, squamous cell carcinoma of the head and neck, urothelial cancer, endometrial cancer, NSCLC, and gastric or gastroesophageal junction adenocarcinoma. The expansion cohorts are limited to the following tumor types: endometrial, SCCHN, CRC, and tumors with an activating mutation in PIK3Ca.
2. Subjects must have a tumor that is at least 1 cm in a single dimension and is radiographically apparent on CT or MRI.
3. Eastern Cooperative Oncology Group performance status of 0 or 1 at treatment initiation.
4. Life expectancy estimated to be ≥ 12 weeks
5. Adequate organ and marrow function (subjects must not have received transfusions or growth factor support within 1 month prior to first dose of investigational product) as defined below:

   * Albumin ≥ 3.0 g/dL
   * Hemoglobin ≥ 10.0 g/dL
   * Absolute neutrophil count ≥ 1,000/mm3
   * Platelet count ≥ 100,000/mm3
   * Bilirubin ≤ 1.5 × institutional upper limit of normal (ULN); for subjects with documented/suspected Gilbert's disease, bilirubin should be ≤ 2 × ULN.
   * Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 × ULN; for subjects with liver metastases, AST or ALT ≤ 5 × ULN
   * Creatinine ≤ 1.5×ULN OR calculated creatinine clearance (CrCl) ≥ 60 mL/min for subjects with creatinine levels > 1.5× ULN.

Subjects who meet any of the following exclusion criteria will not be eligible to receive investigational product:

1. Concurrent enrollment in another clinical study, unless it is an observational (non interventional) clinical study, a specimen-collection study or the follow-up period of an interventional study.
2. Received more than 4 doses of nonsteroidal anti-inflammatory drugs or COX-2 inhibitors within 2 weeks prior to study treatment initiation.
3. History of allergy or hypersensitivity, GI bleed, or ulceration secondary to nonsteroidal anti-inflammatory drugs or COX-2 inhibitors.
4. History of GI ulcer within 1 year of treatment initiation or history of untreated helicobacter pylori infection. Subjects with history of treated helicobacter pylori infection with confirmation of eradication are eligible
5. History of diverticulitis or any GI bleed within 2 years of treatment initiation.
6. Receipt of any anticancer therapy within the following windows:

   * Small molecule tyrosine kinase inhibitor (TKI) therapy (including investigational) within 2 weeks or 5 half-lives prior to treatment initiation, whichever is longer
   * Any type of anti-cancer antibody or cytotoxic chemotherapy within 4 weeks prior to treatment initiation
   * Radiation therapy for bone metastasis within 2 weeks, any other external radiation therapy within 4 weeks before treatment initiation. Patients with clinically relevant ongoing complications from prior radiation therapy are not eligible
   * Other investigational therapy within 2 weeks or 5 half-lives prior to dosing, whichever is longer
7. Subjects with active or untreated central nervous system (CNS) metastases
8. New York Heart Association Classification II, III or IV.
9. Baseline QTcF > 470 milliseconds
10. Receipt of live attenuated vaccines within 30 days prior to the first dose of investigational product. (Killed virus or other non-live vaccines are allowed (including most seasonal influenza vaccines, streptococcus pneumonia vaccines, and newly approved COVID-19 vaccines).
11. Active autoimmune disease or inflammatory disorders including inflammatory bowel disease (e.g., ulcerative colitis or Crohn's disease) requiring systemic treatment (i.e., with use of disease modifying agents, systemic corticosteroids or immunosuppressive drug) within 2 years prior to treatment initiation.
12. Known human immunodeficiency virus (HIV) infection, active Hepatitis B (HBV), or hepatitis C (HCV). Active HBV is defined as a known positive HBsAg result. Active HCV is defined by a known positive HCV antibody result and known quantitative HCV RNA results greater than the lower limits of detection of the assay. Patients receiving antiviral therapy for Hepatitis B or C also are not eligible
13. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations including a history of substance abuse that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent.
14. Subjects who are receiving anti-coagulant therapy or who are considered to be at increased risk of bleeding (i.e bleeding disorder or coagulopathy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2020-05-06 (Actual); Primary Completion 2024-09-25 (Actual); Study Completion 2024-09-25 (Actual)

PRIMARY OUTCOMES:
Determination of maximum tolerated dose and/or recommended Phase 2 dose (RP2D) and optimum dose schedule for TPST-1495 as a single agent and in combination with pembrolizumab | From start of treatment to treatment termination visit, up to 24 months
  Determination of maximum tolerated dose and/or recommended Phase 2 dose (RP2D) and optimum dose schedule for TPST-1495 as a single agent and in combination with pembrolizumab based on dose limiting toxicities

SECONDARY OUTCOMES:
Incidence of adverse events and serious adverse events as assessed by NCI-CTCAE v.5.0 | From start of treatment to treatment termination visit, up to 24 months
  Incidence of treatment-emergent adverse events and serious adverse events for TPST-1495
Assess pharmacokinetics: maximum serum concentration (Cmax) | From start of treatment to treatment termination visit, up to 24 months
  Maximum serum concentration (Cmax) of TPST-1495
Assess pharmacokinetics: area under the serum concentration-time curve (AUC) | From start of treatment to treatment termination visit, up to 24 months
  Area under the serum concentration-time curve (AUC) of TPST-1495
Assess pharmacokinetics: Clearance (CL) | From start of treatment to treatment termination visit, up to 24 months
  Clearance (CL) of TPST-1495
Assess pharmacokinetics: terminal elimination half-life (t 1/2) | From start of treatment to treatment termination visit, up to 24 months
  Terminal elimination half-life (t 1/2) of TPST-1495
Overall response rate (ORR) using RECIST version 1.1 | From start of treatment to treatment termination visit, up to 24 months
  Preliminary efficacy of TPST-1495 as a single agent and in combination with pembrolizumab as assessed by overall response rate (ORR) using RECIST version 1.1
Progression free survival (PFS) | From start of treatment to treatment termination visit, up to 24 months
  Preliminary efficacy of TPST-1495 as a single agent and in combination with pembrolizumab as assessed by progression free survival (PFS)
Duration of response (DoR) | From start of treatment to treatment termination visit, up to 24 months
  Preliminary efficacy of TPST-1495 as a single agent and in combination with pembrolizumab as assessed by duration of response (DoR)

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Whiting, MD PhD, Study Director — Tempest Therapeutics
Locations (11):
- United States (11):
  - University of Colorado, Aurora, Colorado
  - Sidney Kimmel Cancer Center, Johns Hopkins School of Medicine, Baltimore, Maryland
  - Baystate Gynecologic Oncology, Springfield, Massachusetts
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - START Midwest, Grand Rapids, Michigan
  - Carolina BioOncology Institute, Huntersville, North Carolina
  - SCRI-OK Stephenson Cancer Center, Oklahoma City, Oklahoma
  - University of Pennsylvania Perelman School of Medicine, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Tennessee Oncology, Nashville, Tennessee
  - South Texas Accelerated Research Therapeutics (START), San Antonio, Texas

REFERENCES:
- [Derived] Wang D, Cabalag CS, Clemons NJ, DuBois RN. Cyclooxygenases and Prostaglandins in Tumor Immunology and Microenvironment of Gastrointestinal Cancer. Gastroenterology. 2021 Dec;161(6):1813-1829. doi: 10.1053/j.gastro.2021.09.059. Epub 2021 Oct 2. PMID 34606846